CLINICAL TRIAL: NCT03109145
Title: MyHealtheVet to Enable Shared Decision Making Regarding Menopausal and Associated Symptoms in Postmenopausal Women Veterans
Brief Title: MyHealtheVet to Enable Shared Decision Making Regarding Menopausal in Postmenopausal Women Veterans (MEANS)
Acronym: MEANS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miami VA Healthcare System (U.S. Federal Agency)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Stuti Dang, Physician, Miami VA Healthcare System
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pfizer-MEANS; 15911255 (Other Grant/Funding Number: Pfizer)
Record Dates: First submitted 2016-12-12; First posted 2017-04-12 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Menopause
Keywords: Shared decision making; Knowledge; Patient portal; Secure messaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Menopause educational secure messaging (Experimental): Secure messages that provide information about menopause and treatment option for menopause symptoms.
  Interventions: Other: Menopause educational secure messaging
- Usual care: Control (No Intervention): Control group of eligible women patients between 45-60 years who do not receive the intervention at the West Palm Beach and Orlando Veterans Healthcare System. Usual care participants did not receive the educational secure messages.

INTERVENTIONS:
Other: Menopause educational secure messaging — Participants read educational material about menopause and treatment option for menopause symptoms once a week using secure messaging on a electronic patient portal.
  Arms: Menopause educational secure messaging

SUMMARY:
The purpose of this research study is to examine the impact of educational secure messages on menopause. In particular, the investigators will examine whether the secure messages increase menopause knowledge and communication between patients and their providers.

DETAILED DESCRIPTION:
The overall goal of this project is to determine the effectiveness of the MEANS (MyHealtheVet to Enable And Negotiate for Shared decision making) intervention in improving women's self-reported knowledge and rates of diagnosis and appropriate management of menopause symptoms. The proposed intervention is an educational and shared decision making platform for menopause symptoms to improve communication between patients and their providers regarding menopause symptoms. MEANS combines educational secure messages through the Veterans Affairs online Personal Health Record called MyHealtheVet, along with face-to-face and print interventions.

MEANS will be applied in target population consisting of postmenopausal women Veterans ages 45 to 60 who receive primary care at the Miami Veterans Affairs Healthcare System. This project will enroll women in MyHealtheVet, develop a library of menopause symptoms material for distribution, and evaluate how useful of MyHealtheVet use for educating and tracking women regarding menopause symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Women Veterans, age 45-60
* Receive primary care at the Miami Veterans Affairs Healthcare System
* Able to communicate in English
* Already or willing to register and become authenticated in the patient health portal, MyHealtheVet.
* Able to use read, understand, and respond to secure messages using patient health portal.

Exclusion Criteria:

* Not willing to register and become authenticated for patient health portal.
* Not willing to receive educational secure messages from patient health portal.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 859 (Actual)
Dates: Start 2014-10; Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Menopause Knowledge | 6-months
  Total menopause knowledge score (a) before and after the intervention, an average of 6-months and (b) compared to a control group of eligible women patients between 45-60 years who do not receive the intervention at the West Palm Beach and Orlando Veterans Healthcare System. Score is the percent of knowledge questions answered correctly (0 - 100%)
Feasibility of patient portal use for educating and tracking women regarding menopause and menopause related symptoms. | 6-months
  The study will send weekly secure messages regarding menopause, and ask participants to report their menopause related symptoms by secure messaging. The research study will track the number of times participants read the weekly information sent via MyHealtheVet and the proportion of times they respond.

SECONDARY OUTCOMES:
Shared decision making | Through study completion, an average of 3-years
  Self-reported rate of shared decision making among women veteran and their providers.
Menopause related diagnosis | Through study completion, an average of 3-years
  Rates of diagnosis and appropriate management of menopause related symptoms and use of hormone therapy.
Focus Group | 6-months
  Qualitative assessment of the interventions through participant semi-structure focus group interviews.
Patient portal registration and authentication | Through study completion, an average of 3-years
  Measure the number of eligible women patients in the Miami Veterans Healthcare System who are enrolled and authenticated in the patient portal before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Stuti Dang, MD, MPH, Principal Investigator — Miami VA Healthcare System
Locations (1):
- Miami Veterans Affairs Healthcare System, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lamba AH, Muralidhar K, Jain A, Tang F, Gomez-Marin O, Levis S, Dang S. Characteristics of Women Enrolled in a Patient Portal Intervention for Menopause. Womens Health Rep (New Rochelle). 2020 Oct 26;1(1):500-510. doi: 10.1089/whr.2020.0091. eCollection 2020. PMID 33786517
- [Derived] Dang S, Thavalathil B, Ruiz D, Gomez-Orozco C, Gomez-Marin O, Levis S. A Patient Portal Intervention for Menopause Knowledge and Shared Decision-Making. J Womens Health (Larchmt). 2019 Dec;28(12):1614-1622. doi: 10.1089/jwh.2018.7461. Epub 2019 Aug 7. PMID 31390282